CLINICAL TRIAL: NCT07340996
Title: Effects of Beta Caryophyllene Supplementation on Autonomic Regulation and Apnea Performance in Elite Divers - a Randomized Crossover Trial
Brief Title: Beta Caryophyllene & Apnea Performance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chih-Hui Chiu (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor-Investigator, Chih-Hui Chiu, Professor, National Taiwan Sport University
Organization: National Taiwan Sport University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 115-1; 115-1 (Other: NTUS)
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: EXERCISE PERFORMANCE
Keywords: freediving
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: randomized crossover design with double-blind methodology
Who Masked: Investigator
Masking Description: placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): supplementation β-caryophyllene
  Interventions: Dietary Supplement: interventions; Dietary Supplement: Placebo
- placebo (Placebo Comparator): placebo
  Interventions: Dietary Supplement: interventions; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: interventions — supplementation of β-caryophyllene
Dietary Supplement: Placebo — Participants consumed placebo capsules (PLA trial)

SUMMARY:
The purpose of this study is to investigate whether β-caryophyllene supplementation can enhance the static apnea capacity of freedivers.

DETAILED DESCRIPTION:
Using a randomized crossover design with double-blind methodology, participants were assigned to either the β-caryophyllene trial (BCP) trial or the placebo (PLA) trial, which without β-caryophyllene. Participants consumed either 200 mg of β-caryophyllene capsules (BCP trial) or placebo capsules (PLA trial) based on pre-test results. After a 30-minute rest period and warm-up, a single maximal voluntary static breath-hold test was conducted. Breath-hold duration and physiological and salivary biochemical indicators before and after the breath-hold test were observed.

ELIGIBILITY:
Inclusion Criteria:

* With over 3 years of freediving experience

Exclusion Criteria:

* Without over 3 years of freediving experience

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male subjects
Enrollment: 15 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Breath-hold duration | 30 minutes after intervention
  Measure the duration of static breath-holding

CONTACTS AND LOCATIONS:
Overall Officials: Chih Hui Chiu, Principal Investigator — National Taiwan University of Sport
Locations (1):
- National Taiwan University of Sport, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2026-01-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT07340996/Prot_000.pdf